CLINICAL TRIAL: NCT04640194
Title: The TRISTARDS Trial - ThRombolysIS Therapy for ARDS A Phase IIb/III Operationally Seamless, Open-label, Randomised, Sequential, Parallel-group Adaptive Study to Evaluate the Efficacy and Safety of Daily Intravenous Alteplase Treatment Given up to 5 Days on Top of Standard of Care (SOC) Compared With SOC Alone, in Patients With Acute Respiratory Distress Syndrome (ARDS) Triggered by COVID-19
Brief Title: A Study to Test Whether Different Doses of Alteplase Help People With Severe Breathing Problems Because of COVID-19
Acronym: TRISTARDS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0135-0347; 2020-002913-16 (EudraCT Number)
Record Dates: First submitted 2020-11-20; First posted 2020-11-23 (Actual); Results first posted 2024-03-07 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Standard of Care; Tissue Plasminogen Activator

STUDY DESIGN:
Intervention Model Description: The study comprises two parts: Part 1 (dose-finding, Phase IIb) and Part 2 (confirmatory, Phase III)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Part 1: Alteplase low dose (Experimental): 0.3 milligram/kilogram (mg/kg) over 2 hours (Day 1) immediately followed by daily infusion of 0.02 mg/kg/hour over 12 hours (starting on Day 1 and up to Day 5), plus Standard of Care (SOC). One optional additional infusion of 0.3 mg/kg over 2 hours could be given once on Days 2 to 5 in case of clinical worsening, per investigator judgement. Part 1 subjects were randomized equally (1:1:1) across the three Part 1 arms.
  Interventions: Procedure: Standard of care; Drug: Alteplase low dose
- Part 1: Alteplase high dose (Experimental): 0.6 milligram/kilogram (mg/kg) over 2 hours (Day 1) immediately followed by daily infusion of 0.04 mg/kg/hour over 12 hours (starting on Day 1 and up to Day 5), plus Standard of Care (SOC). One optional additional infusion of 0.6 mg/kg over 2 hours could be given once on Days 2 to 5 in case of clinical worsening, per investigator judgement. Part 1 subjects were randomized equally (1:1:1) across the three Part 1 arms.
  Interventions: Procedure: Standard of care; Drug: Alteplase high dose
- Part 1: Standard of Care (Other): Standard of Care included best possible treatment regimen established locally and was in line with current guidelines for Acute respiratory distress syndrome treatment. Part 1 subjects were randomized equally (1:1:1) across the three Part 1 arms.
  Interventions: Procedure: Standard of care
- Part 2: Alteplase high dose - non-invasive mechanical ventilation (NIV) patients (Experimental): 0.6 milligram/kilogram (mg/kg) over 2 hours (Day 1) immediately followed by daily infusion of 0.04 mg/kg/hour over 12 hours (starting on Day 1 and up to Day 5), plus Standard of Care (SOC). One optional additional infusion of 0.6 mg/kg over 2 hours could be given once on Days 2 to 5 in case of clinical worsening, per investigator judgement. Non-invasive mechanical ventilation (NIV) patients are those with a baseline World Health Organization (WHO) Clinical Progression Scale value of 6. Part 2 subjects were randomized 2 (Alteplase) to 1 (SOC).
  Interventions: Procedure: Standard of care; Drug: Alteplase high dose
- Part 2: Standard of Care - non-invasive mechanical ventilation (NIV) patients (Other): Standard of Care included best possible treatment regimen established locally and was in line with current guidelines for Acute respiratory distress syndrome treatment. Non-invasive mechanical ventilation (NIV) patients are those with a baseline World Health Organization (WHO) Clinical Progression Scale value of 6. Part 2 subjects were randomized 2 (Alteplase) to 1 (SOC).
  Interventions: Procedure: Standard of care
- Part 2: Alteplase high dose - invasive mechanical ventilation (IMV) patients (Experimental): 0.6 milligram/kilogram (mg/kg) over 2 hours (Day 1) immediately followed by daily infusion of 0.04 mg/kg/hour over 12 hours (starting on Day 1 and up to Day 5), plus Standard of Care (SOC). One optional additional infusion of 0.6 mg/kg over 2 hours could be given once on Days 2 to 5 in case of clinical worsening, per investigator judgement. Invasive mechanical ventilation (IMV) patients are those with a baseline World Health Organization (WHO) Clinical Progression Scale value of 7, 8 or 9. Part 2 subjects were randomized 2 (Alteplase) to 1 (SOC).
  Interventions: Procedure: Standard of care; Drug: Alteplase high dose
- Part 2: Standard of Care - invasive mechanical ventilation (IMV) patients (Other): Standard of Care included best possible treatment regimen established locally and was in line with current guidelines for Acute respiratory distress syndrome treatment. Invasive mechanical ventilation (IMV) patients are those with a baseline World Health Organization (WHO) Clinical Progression Scale value of 7, 8 or 9. Part 2 subjects were randomized 2 (Alteplase) to 1 (SOC).
  Interventions: Procedure: Standard of care

INTERVENTIONS:
Procedure: Standard of care — Standard of Care (SOC) includes any supportive measures applied in hospital, specifically on an intensive care unit (ICU), such as for example the use of non-invasive or invasive ventilation, oxygen masks, haemodynamic support, if needed, sedation, as well as medical therapies commonly used in patients suffering from acute respiratory distress syndrome (ARDS) or its complications. SOC should include best possible treatment regimen established locally and should be in line with current guidelines for ARDS treatment.
Drug: Alteplase low dose — 0.3 milligram/kilogram (mg/kg) over 2 hours (Day 1) immediately followed by daily infusion of 0.02 mg/kg/hour over 12 hours (starting on Day 1 and up to Day 5). One optional additional infusion of 0.3 mg/kg over 2 hours could be given once on Days 2 to 5 in case of clinical worsening, per investigator judgement.
  Arms: Part 1: Alteplase low dose
Drug: Alteplase high dose — 0.6 milligram/kilogram (mg/kg) over 2 hours (Day 1) immediately followed by daily infusion of 0.04 mg/kg/hour over 12 hours (starting on Day 1 and up to Day 5). One optional additional infusion of 0.6 mg/kg over 2 hours could be given once on Days 2 to 5 in case of clinical worsening, per investigator judgement.
  Arms: Part 1: Alteplase high dose; Part 2: Alteplase high dose - invasive mechanical ventilation (IMV) patients; Part 2: Alteplase high dose - non-invasive mechanical ventilation (NIV) patients

SUMMARY:
This is a study in adults with severe breathing problems because of COVID-19. People who are in hospital on breathing support can participate in the study. The purpose of the study is to find out whether a medicine called alteplase helps people get better faster.

The study has 2 parts. In the first part, participants are put into 3 groups by chance. Participants in 2 of the groups get 2 different doses of alteplase, in addition to standard treatment.

Participants in the third group get standard treatment. In the second part of the study, participants are put into 2 groups by chance. One group gets alteplase and standard treatment. The other group gets only standard treatment. Alteplase is given as an infusion into a vein. In both study parts, treatments are given for 5 days. Doctors monitor patients and check whether their breathing problems improve. They compare results between the groups after 1 month.

Participants are in the study for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years (or above legal age, e.g. UK ≥16 years)
* ARDS with PaO2*/FiO2 ratio >100 and ≤300, either on non-invasive ventilator support, OR on mechanical ventilation (<48 hours since intubation),

  * with bilateral opacities in chest X-ray or CT scan (not fully explained by effusions, lobar/lung collapse, or nodules)
  * with respiratory failure (not fully explained by cardiac failure/fluid overload) (*or estimation of PaO2/FiO2 from pulse oximetry (SpO2/FiO2))
* SARS-CoV-2 positive (laboratory-confirmed reverse transcription polymerase chain reaction (RT PCR) test)
* Fibrinogen level ≥ lower limit of normal (according to local laboratory)
* D-Dimer ≥ upper limit of normal (ULN) according to local laboratory
* Signed and dated written informed consent in accordance with ICH Good Clinical Practice (GCP) and local legislation prior to admission to the Trial

Exclusion Criteria:

* Massive confirmed pulmonary embolism (PE) with haemodynamic instability at trial entry, or any (suspected or confirmed) PE that is expected to require therapeutic dosages of anticoagulants during the treatment period
* Indication for therapeutic dosages of anticoagulants at trial entry
* Patients on mechanical ventilation for longer than 48 hours
* Chronic pulmonary disease i.e. with known forced expiratory volume in 1 second (FEV1) <50%, requiring home oxygen, or oral steroid therapy or hospitalisation for exacerbation within 12 months, or significant chronic pulmonary disease in the Investigator's opinion, or primary pulmonary arterial hypertension
* Has a Do-Not-Intubate (DNI) or Do-Not-Resuscitate (DNR) order
* In the opinion of the investigator not expected to survive for > 48 hours after admission
* Planned interventions during the first 5 days after randomisation, such as surgery, insertion of central catheter or arterial line, drains, etc.
* Patients with known hypersensitivity to the active substance alteplase, gentamicin (a trace residue from the manufacturing process) or to any of the excipients
* Significant bleeding disorder at present or within the past 3 months, known haemorrhagic diathesis
* Patients receiving effective oral anticoagulant treatment, e.g. vitamin K antagonists with International normalised ratio (INR) >1.3, or any direct oral anticoagulant within the past 48 hours Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2022-07-19 (Actual); Study Completion 2022-07-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (37):
- Austria (2):
  - LKH Klagenfurt am Woerthersee, Klagenfurt
  - Wiener Gesundheitsverbund Klinik Favoriten, Vienna
- Belgium (3):
  - ULB Hopital Erasme, Brussels
  - Centre Hospitalier Universitaire de Liège, Liège
  - Ottignies - HOSP St-Pierre, Ottignies
- Hospital Mae de Deus, Porto Alegre, Brazil
- France (8):
  - HOP Bicêtre, Le Kremlin-Bicêtre
  - HOP Roger Salengro, Lille
  - HOP Melun-Sénart, Melun
  - HOP Hôtel-Dieu, Nantes
  - HOP Cochin, Paris
  - HOP Européen G. Pompidou, Paris
  - HOP Robert Debré, Reims
  - HOP Civil, Strasbourg
- Germany (6):
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Leipzig, Leipzig
  - Universitätsklinikum Mannheim GmbH, Mannheim
  - Klinikum der Universität München - Campus Großhadern, München
  - Petrus-Krankenhaus, Wuppertal
- King George Hospital, Visakhapatnam, India
- Italy (2):
  - IRCCS San Raffaele, Milan
  - Istituto Clinico Humanitas, Rozzano (MI)
- Hospital Miri, Miri, Malaysia
- Hospital Cardiologica Aguascalientes, Aguascalientes, Mexico
- Netherlands (3):
  - Gelre Ziekenhuizen Apeldoorn, Apeldoorn
  - Rijnstate Hospital, Arnhem
  - Canisius-Wilhelmina ziekenhuis, Nijmegen
- Russia (4):
  - City Clinical Hospital # 40 of the Moscow Health Department, Moscow
  - Moscow 1st State Med.Univ.n.a.I.M.Sechenov, Moscow
  - City Clinical Emergency Hospital, Ryazan
  - State Budget Institution of Healthcare Leningradskaya region "Kirovskaya Interdistrict Hospital", Saint Petersburg
- Spain (4):
  - Hospital del Mar, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Puerta del Mar, Cadiz
  - CS Parc Taulí, Sabadell
- Izmir Dr. Suat Seren Gogus Hastaliklari ve Cerrahisi Egitim ve Arastirma Hastanesi, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
  The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Landoni G, Chowdary P, Meziani F, Creteur J, De Schryver N, Motsch J, Henrichmoeller I, Pages A, Peter N, Danays T, Weigand MA; TRISTARDS Investigators. Alteplase in COVID-19 severe hypoxemic respiratory failure: the TRISTARDS multicenter randomized trial. Ann Intensive Care. 2024 Nov 10;14(1):170. doi: 10.1186/s13613-024-01386-z. PMID 39522090
- See also: Related Info — https://www.mystudywindow.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A Phase IIb/III randomised, controlled, open-label, sequential, parallel-group, operationally seamless adaptive study with two parts. Part 1 was a Phase IIb proof-of-concept exploratory comparison of two groups each receiving a different dose of alteplase plus Standard of Care (SOC) versus a group receiving SOC alone. Part 2 was a confirmatory Phase III study; Part 2 will include one group receiving the selected dose of alteplase plus SOC vs. one group receiving SOC alone.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Overall Study
Arm/Group | Part 1: Alteplase Low Dose | Part 1: Alteplase High Dose | Part 1: Standard of Care | Part 2: Alteplase High Dose - Non-invasive Mechanical Ventilation (NIV) Patients | Part 2: Standard of Care - Non-invasive Mechanical Ventilation (NIV) Patients | Part 2: Alteplase High Dose - Invasive Mechanical Ventilation (IMV) Patients | Part 2: Standard of Care - Invasive Mechanical Ventilation (IMV) Patients
Started | 20 | 20 | 22 | 17 | 8 | 12 | 5
Completed (Completed treatment) | 17 | 12 | 22 | 9 | 8 | 8 | 5
Not Completed | 3 | 8 | 0 | 8 | 0 | 4 | 0
Not completed — Adverse Event | 3 | 7 | 0 | 5 | 0 | 4 | 0
Not completed — pO2/FIO2 ratio too high | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — fibrinogen level too low | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — mild bleeding | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Transferred from Intensive Care Unit to Hospital Ward | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) consisted of all randomised patients with at least one baseline and one post baseline assessment relating to the primary endpoint of interest.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Alteplase Low Dose | Part 1: Alteplase High Dose | Part 1: Standard of Care | Part 2: Alteplase High Dose - Non-invasive Mechanical Ventilation (NIV) Patients | Part 2: Standard of Care - Non-invasive Mechanical Ventilation (NIV) Patients | Part 2: Alteplase High Dose - Invasive Mechanical Ventilation (IMV) Patients | Part 2: Standard of Care - Invasive Mechanical Ventilation (IMV) Patients | Total
Number analyzed (Participants) | 20 | 20 | 22 | 17 | 8 | 12 | 5 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (12.0) | 61.6 (9.8) | 60.3 (13.0) | 63.4 (11.5) | 60.5 (10.9) | 59.7 (11.1) | 67.6 (10.5) | 61.5 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 3 | 9 | 3 | 5 | 1 | 1 | 32
  Male | 10 | 17 | 13 | 14 | 3 | 11 | 4 | 72
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 13 | 13 | 14 | 10 | 3 | 7 | 1 | 61
  Native Hawaiian or Other Pacific Islander & White | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  American Indian or Alaska Native & White | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Missing | 7 | 7 | 5 | 5 | 5 | 5 | 4 | 38
WHO Clinical Progression Scale [Count of Participants; unit: Participants] — World Health Organization (WHO) Clinical Progression Scale ranges from 0 to 10, low score indicates better outcome. 0=Uninfected; no viral RNA detected 1=Asymptomatic; viral RNA detected 2=Symptomatic; independent 3=Symptomatic; assistance needed 4=Hospitalised; no oxygen therapy 5=Hospitalised; oxygen by mask or nasal prongs 6=Hospitalised; oxygen by NIV or high flow 7=Intubation and mechanical ventilation, PaO2/FiO2=150 or SpO2/FiO2=200 8=Mechanical ventilation PaO2/FiO2 <150 (SpO2/FiO2 <200) or vasopressors 9=Mechanical ventilation PaO2/FiO2 <150 and vasopressors, dialysis, or ECMO 10=Dead.
  Participants
    0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    6 | 16 | 16 | 16 | 17 | 8 | 0 | 0 | 73
    7 | 1 | 1 | 3 | 0 | 0 | 1 | 3 | 9
    8 | 2 | 0 | 1 | 0 | 0 | 8 | 0 | 11
    9 | 1 | 3 | 2 | 0 | 0 | 3 | 2 | 11
    10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to Clinical Improvement or Hospital Discharge up to Day 28
Description: From randomisation to either an improvement of 2 points on the 11-point World Health Organization (WHO) Clinical Progression Scale (from 0 to 10, a low score indicates a better outcome) or discharge from the hospital, whichever comes first. Full scale:
  0=Uninfected; no viral RNA detected
  1. Asymptomatic; viral RNA detected
  2. Symptomatic; independent
  3. Symptomatic; assistance needed
  4. Hospitalised; no oxygen therapy
  5. Hospitalised; oxygen by mask or nasal prongs
  6. Hospitalised; oxygen by NIV or high flow
  7. Intubation and mechanical ventilation, PaO2/FiO2=150 or SpO2/FiO2=200
  8. Mechanical ventilation PaO2/FiO2<150 (SpO2/FiO2<200) or vasopressors
  9. Mechanical ventilation PaO2/FiO2<150 and vasopressors, dialysis, or ECMO
  10. Dead
  Patients that have not met the endpoint were censored at Day 28 if they died prior to Day 28. Patients receiving bail out therapy without having first met the endpoint, were censored on the day of bail-out (hypothetical estimand).
Time Frame: Up to 28 days.
Population: Full Analysis Set (FAS) consisted of all randomised patients with at least one baseline and one post baseline assessment relating to the primary endpoint.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Part 1: Alteplase Low Dose | Part 1: Alteplase High Dose | Part 1: Standard of Care | Part 2: Alteplase High Dose - Non-invasive Mechanical Ventilation (NIV) Patients | Part 2: Standard of Care - Non-invasive Mechanical Ventilation (NIV) Patients | Part 2: Alteplase High Dose - Invasive Mechanical Ventilation (IMV) Patients | Part 2: Standard of Care - Invasive Mechanical Ventilation (IMV) Patients
Number analyzed (Participants) | 20 | 20 | 22 | 17 | 8 | 12 | 5
days | NA [14.0 to NA] — Median and Upper limit was not achieved, due to insufficient numbers of participants with events. | 19.0 [9.0 to NA] — Upper limit was not achieved, due to insufficient numbers of participants with events. | NA [17.0 to NA] — Median and Upper limit was not achieved, due to insufficient numbers of participants with events. | 22.0 [7.0 to NA] — Upper limit was not achieved, due to insufficient numbers of participants with events. | NA [8.0 to NA] — Median and Upper limit was not achieved, due to insufficient numbers of participants with events. | 25.5 [13.0 to NA] — Upper limit was not achieved, due to insufficient numbers of participants with events. | NA [4.0 to NA] — Median and Upper limit was not achieved, due to insufficient numbers of participants with events.
Statistical Analysis 1: Comparison: Part 1: Alteplase Low Dose vs Part 1: Standard of Care; Unadjusted Hazard Ratio: Cox proportional hazard model containing fixed effect for treatment. The confidence intervals was determined using the Wald method to determine the variance; Test type: Other; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.39 to 2.61] — A hazard ratio > 1 favours the alteplase dose group over standard of care alone
Statistical Analysis 2: Comparison: Part 1: Alteplase Low Dose vs Part 1: Standard of Care; Adjusted Hazard Ratio: Cox proportional hazard model containing fixed effect for treatment,ventilation status at baseline and age. The confidence intervals was determined using the Wald method to determine the variance; Test type: Other; Hazard Ratio (HR) = 1.23, 95% CI 2-sided [0.46 to 3.27] — A hazard ratio > 1 favours the alteplase dose group over standard of care alone
Statistical Analysis 3: Comparison: Part 1: Alteplase High Dose vs Part 1: Standard of Care; [analysis description as in outcome 1, analysis 1]; Test type: Other; Hazard Ratio (HR) = 1.75, 95% CI 2-sided [0.73 to 4.15] — A hazard ratio > 1 favours the alteplase dose group over standard of care alone
Statistical Analysis 4: Comparison: Part 1: Alteplase High Dose vs Part 1: Standard of Care; [analysis description as in outcome 1, analysis 2]; Test type: Other; Hazard Ratio (HR) = 2.04, 95% CI 2-sided [0.83 to 5.01] — A hazard ratio > 1 favours the alteplase dose group over standard of care alone
Statistical Analysis 5: Comparison: Part 2: Alteplase High Dose - Non-invasive Mechanical Ventilation (NIV) Patients vs Part 2: Standard of Care - Non-invasive Mechanical Ventilation (NIV) Patients; [analysis description as in outcome 1, analysis 1]; Test type: Other; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.35 to 3.66] — A hazard ratio > 1 favours the alteplase dose group over standard of care alone
Statistical Analysis 6: Comparison: Part 2: Alteplase High Dose - Non-invasive Mechanical Ventilation (NIV) Patients vs Part 2: Standard of Care - Non-invasive Mechanical Ventilation (NIV) Patients; [analysis description as in outcome 1, analysis 2]; Test type: Other; Hazard Ratio (HR) = 1.19, 95% CI 2-sided [0.33 to 4.22] — A hazard ratio > 1 favours the alteplase dose group over standard of care alone

2. Secondary Outcome: Number of Subjects With Major Bleeding Events (MBE) at Day 6
Description: Number of subjects with major bleeding events (MBE). Major bleeding events (MBE) according to International Society on Thrombosis and Haemostasis [ISTH] definition until Day 6. Definition of a major bleed:
  •Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intra-articular or pericardial, or intramuscular with compartment syndrome,
  and/or
  •Bleeding associated with a reduction in hemoglobin of at least 2 gram/deciliter (1.24 millimole/Liter), or leading to transfusion of two or more units of blood or packed cells
  and/or
  •Fatal bleed
Time Frame: From start of treatment (Alteplase) or randomisation (SOC) (day 1) till Day 6, up to 6 days.
Population: The Treated Set (TS) consisted of all patients who were randomised and, for patients in the alteplase groups, treated with at least one dose of trial drug.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: Alteplase Low Dose: 0.3 milligram/kilogram (mg/kg) over 2 hours (Day 1) immediately followed by daily infusion of 0.02 mg/kg/hour over 12 hours (starting on Day 1 and up to Day 5), plus Standard of Care (SOC). One optional additional infusion of 0.3 mg/kg over 2 hours could be given once on Days 2 to 5 in case of clinical worsening, per investigator judgement.
- Part 1: Alteplase High Dose: 0.6 milligram/kilogram (mg/kg) over 2 hours (Day 1) immediately followed by daily infusion of 0.04 mg/kg/hour over 12 hours (starting on Day 1 and up to Day 5), plus Standard of Care (SOC). One optional additional infusion of 0.6 mg/kg over 2 hours could be given once on Days 2 to 5 in case of clinical worsening, per investigator judgement.
- Part 1: Standard of Care: Standard of Care included best possible treatment regimen established locally and was in line with current guidelines for Acute respiratory distress syndrome treatment.
- Part 2: Alteplase High Dose - Non-invasive Mechanical Ventilation (NIV) Patients: 0.6 milligram/kilogram (mg/kg) over 2 hours (Day 1) immediately followed by daily infusion of 0.04 mg/kg/hour over 12 hours (starting on Day 1 and up to Day 5), plus Standard of Care (SOC). One optional additional infusion of 0.6 mg/kg over 2 hours could be given once on Days 2 to 5 in case of clinical worsening, per investigator judgement. Non-invasive mechanical ventilation (NIV) patients are those with a baseline World Health Organization (WHO) Clinical Progression Scale value of 6.
- Part 2: Standard of Care - Non-invasive Mechanical Ventilation (NIV) Patients: Standard of Care included best possible treatment regimen established locally and was in line with current guidelines for Acute respiratory distress syndrome treatment. Non-invasive mechanical ventilation (NIV) patients are those with a baseline World Health Organization (WHO) Clinical Progression Scale value of 6.
- Part 2: Alteplase High Dose - Invasive Mechanical Ventilation (IMV) Patients: 0.6 milligram/kilogram (mg/kg) over 2 hours (Day 1) immediately followed by daily infusion of 0.04 mg/kg/hour over 12 hours (starting on Day 1 and up to Day 5), plus Standard of Care (SOC). One optional additional infusion of 0.6 mg/kg over 2 hours could be given once on Days 2 to 5 in case of clinical worsening, per investigator judgement. Invasive mechanical ventilation (IMV) patients are those with a baseline World Health Organization (WHO) Clinical Progression Scale value of 7, 8 or 9.
- Part 2: Standard of Care - Invasive Mechanical Ventilation (IMV) Patients: Standard of Care included best possible treatment regimen established locally and was in line with current guidelines for Acute respiratory distress syndrome treatment. Invasive mechanical ventilation (IMV) patients are those with a baseline World Health Organization (WHO) Clinical Progression Scale value of 7, 8 or 9.
Arm/Group | Part 1: Alteplase Low Dose | Part 1: Alteplase High Dose | Part 1: Standard of Care | Part 2: Alteplase High Dose - Non-invasive Mechanical Ventilation (NIV) Patients | Part 2: Standard of Care - Non-invasive Mechanical Ventilation (NIV) Patients | Part 2: Alteplase High Dose - Invasive Mechanical Ventilation (IMV) Patients | Part 2: Standard of Care - Invasive Mechanical Ventilation (IMV) Patients
Number analyzed (Participants) | 20 | 20 | 22 | 17 | 8 | 12 | 5
Participants | 1 | 4 | 0 | 2 | 0 | 2 | 0
Statistical Analysis 1: Comparison: Part 1: Alteplase Low Dose vs Part 1: Standard of Care; Test type: Other; Risk Difference (RD) = 5.00, 95% CI 2-sided [-10.892 to 24.8734] — Chan and Zhang exact confidence interval
Statistical Analysis 2: Comparison: Part 1: Alteplase High Dose vs Part 1: Standard of Care; Test type: Other; Risk Difference (RD) = 20.00, 95% CI 2-sided [2.3075 to 43.6615] — Chan and Zhang exact confidence interval
Statistical Analysis 3: Comparison: Part 2: Alteplase High Dose - Non-invasive Mechanical Ventilation (NIV) Patients vs Part 2: Standard of Care - Non-invasive Mechanical Ventilation (NIV) Patients; Test type: Other; Risk Difference (RD) = 11.76, 95% CI 2-sided [-24.127 to 36.9012] — Chan and Zhang exact confidence interval

3. Secondary Outcome: All Cause Mortality at Day 28
Description: All cause mortality at Day 28. If it is unknown whether the patient was dead at end of Day 28, then it will be assumed that the patient did not die up to Day 28, regardless of the reason. This unfavorable endpoint is met if:
  * the last known status of the patient is 10 on the WHO clinical progression scale by the end of Day 28, or
  * vital status is dead within 28 days
Time Frame: Up to 28 days.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Alteplase Low Dose | Part 1: Alteplase High Dose | Part 1: Standard of Care | Part 2: Alteplase High Dose - Non-invasive Mechanical Ventilation (NIV) Patients | Part 2: Standard of Care - Non-invasive Mechanical Ventilation (NIV) Patients | Part 2: Alteplase High Dose - Invasive Mechanical Ventilation (IMV) Patients | Part 2: Standard of Care - Invasive Mechanical Ventilation (IMV) Patients
Number analyzed (Participants) | 20 | 20 | 22 | 17 | 8 | 12 | 5
Participants | 2 | 3 | 6 | 1 | 2 | 2 | 2
Statistical Analysis 1: Comparison: Part 1: Alteplase Low Dose vs Part 1: Standard of Care; Adjusted risk difference and 95% confidence interval is based upon average marginal effect Delta method, adjusting for baseline ventilation status, age and treatment; Test type: Other; Risk Difference (RD) = -16.6, 95% CI 2-sided [-38.6 to 5.5] — Calculated as alteplase dose group - standard of care alone
Statistical Analysis 2: Comparison: Part 1: Alteplase High Dose vs Part 1: Standard of Care; [analysis description as in outcome 3, analysis 1]; Test type: Other; Risk Difference (RD) = -11.8, 95% CI 2-sided [-35.1 to 11.6] — Calculated as alteplase dose group - standard of care alone
Statistical Analysis 3: Comparison: Part 2: Alteplase High Dose - Non-invasive Mechanical Ventilation (NIV) Patients vs Part 2: Standard of Care - Non-invasive Mechanical Ventilation (NIV) Patients; Unadjusted risk difference and 95% CI is based upon average marginal effect Delta method, adjusting for treatment; Test type: Other; p = 0.2419, The delta method and average marginal; Risk Difference (RD) = -19.1, 95% CI 2-sided [-51.1 to 12.9] — Calculated as alteplase dose group - standard of care alone

4. Secondary Outcome: Number of Subjects With Treatment Failure at Day 28
Description: Treatment failure defined as all cause mortality or mechanical ventilation at Day 28.
Time Frame: Up to 28 days.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Alteplase Low Dose | Part 1: Alteplase High Dose | Part 1: Standard of Care | Part 2: Alteplase High Dose - Non-invasive Mechanical Ventilation (NIV) Patients | Part 2: Standard of Care - Non-invasive Mechanical Ventilation (NIV) Patients | Part 2: Alteplase High Dose - Invasive Mechanical Ventilation (IMV) Patients | Part 2: Standard of Care - Invasive Mechanical Ventilation (IMV) Patients
Number analyzed (Participants) | 20 | 20 | 22 | 17 | 8 | 12 | 5
Participants | 8 | 8 | 11 | 6 | 3 | 5 | 3
Statistical Analysis 1: Comparison: Part 1: Alteplase Low Dose vs Part 1: Standard of Care; [analysis description as in outcome 3, analysis 1]; Test type: Other; Risk Difference (RD) = -9.0, 95% CI 2-sided [-37.1 to 19.1] — Calculated as alteplase dose group - standard of care alone
Statistical Analysis 2: Comparison: Part 1: Alteplase High Dose vs Part 1: Standard of Care; [analysis description as in outcome 3, analysis 1]; Test type: Other; Risk Difference (RD) = -9.1, 95% CI 2-sided [-37.2 to 19.0] — Calculated as alteplase dose group - standard of care alone
Statistical Analysis 3: Comparison: Part 2: Alteplase High Dose - Non-invasive Mechanical Ventilation (NIV) Patients vs Part 2: Standard of Care - Non-invasive Mechanical Ventilation (NIV) Patients; Adjusted risk difference and 95% CI is based upon average marginal effect Delta method, adjusting for baseline D-dimer status, age, days of NIV support and treatment; Test type: Other; p = 0.2523, The delta method and average marginal; Risk Difference (RD) = 14.5, 95% CI 2-sided [-10.3 to 39.3] — Calculated as alteplase dose group - standard of care alone

5. Secondary Outcome: Number of Ventilator-free Days at Day 28
Description: Number of ventilator-free days (VFDs) from start of treatment to Day 28. 'Ventilator' is defined as 'assisted breathing' but it refers to mechanical invasive ventilation. The number of VFDs starts from when the patient has a 'lasting' value on the WHO clinical progression scale of ≤ 6, and ends on Day 28. A lasting value of ≤ 6 means that the value cannot exceed 6 at a later timepoint. If the patient is liberated from the ventilator on Day x, then the number of VFDs is 28-x. If a patient has withdrawn consent prior to day 28 then he will have a missing value for VFD. In any case, if the status of the patient at Day 28 is death, as determined from the vital status page then the VFD=0.
Time Frame: Up to 28 days.
Population: Full Analysis Set (FAS) consisted of all randomised patients with at least one baseline and one post baseline assessment relating to the primary endpoint. The endpoint was only planned for subjects in Part 1.
Measure: Mean (Standard Error); unit: Days
Arm/Group | Part 1: Alteplase Low Dose | Part 1: Alteplase High Dose | Part 1: Standard of Care
Number analyzed (Participants) | 20 | 20 | 22
Days | 10.6 (2.9) | 11.8 (2.9) | 7.5 (2.7)
Statistical Analysis 1: Comparison: Part 1: Alteplase Low Dose vs Part 1: Standard of Care; Parameters included in model: treatment,ventilation status at baseline, and age; Test type: Other; Mean Difference (Final Values) = 3.1, 95% CI 2-sided [-4.4 to 10.6], Standard Error of Mean 3.7 — Calculated as alteplase dose group - standard of care alone
Statistical Analysis 2: Comparison: Part 1: Alteplase High Dose vs Part 1: Standard of Care; Parameters included in model: treatment,ventilation status at baseline, and age; Test type: Other; Median Difference (Final Values) = 4.3, 95% CI 2-sided [-3.2 to 11.8], Standard Error of Mean 3.7 — Calculated as alteplase dose group - standard of care alone

6. Secondary Outcome: Number of Subjects With Improvement of Sequential (Sepsis-related) Organ Failure Assessment (SOFA) Score by ≥2 Points at Day 6
Description: Number of subjects with improvement of Sequential (sepsis-related) Organ Failure Assessment (SOFA) score by ≥2 points from baseline to end of Day 6. The Sequential Organ Failure Assessment (SOFA) scores six variables: respiratory, coagulation, liver, Cardiovascular, central nervous system and renal. Each variable is score from 0 (best outcome) to 4 (worst outcome) with a total score calculated as the sum of all six variables ranging from 0 (best outcome) to 24 (worst outcome).
Time Frame: Baseline (Day 0) and Day 6 of treatment
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Alteplase Low Dose | Part 1: Alteplase High Dose | Part 1: Standard of Care
Number analyzed (Participants) | 20 | 20 | 22
Participants | 4 | 2 | 6
Statistical Analysis 1: Comparison: Part 1: Alteplase Low Dose vs Part 1: Standard of Care; [analysis description as in outcome 3, analysis 1]; Test type: Other; Risk Difference (RD) = -4.9, 95% CI 2-sided [-29.0 to 19.2] — Calculated as alteplase dose group - standard of care alone
Statistical Analysis 2: Comparison: Part 1: Alteplase High Dose vs Part 1: Standard of Care; [analysis description as in outcome 3, analysis 1]; Test type: Other; Risk Difference (RD) = -15.2, 95% CI 2-sided [-36.8 to 6.3] — Calculated as alteplase dose group - standard of care alone

7. Secondary Outcome: Daily Average PaO2/FiO2 Ratio Change From Baseline to Day 6
Description: Daily average PaO2/FiO2 ratio (or inferred PaO2/FiO2 ratio from SpO2) change from baseline to Day 6. This assessment was measured approximately 3-times daily. All available values on each of these days, regardless of the position of the patient when being measured, were averaged in order to determine the daily average PaO2/FiO2 ratio for that patient. The higher the value the better the health status of the patient. If the patient was still in hospital during day 6 then the day 6 daily average value was used, if available. If the patient was discharged from hospital prior to day 6 then the daily average at the time of hospital discharge was used as a surrogate for day 6, if available. If the patient died prior to day 6 then there was no imputation but the death handled as failure in the determination of the difference in medians and 95% CI. Based upon this, the change from baseline for each patient was calculated.
Time Frame: Up to 6 days.
Population: Full Analysis Set (FAS) consisted of all randomised patients with at least one baseline and one post baseline assessment relating to the primary endpoint. Only subjects with non-missing endpoint data were included. The endpoint was only planned for subjects in Part 1.
Measure: Median (Inter-Quartile Range); unit: PaO2/FiO2 ratio
Arm/Group | Part 1: Alteplase Low Dose | Part 1: Alteplase High Dose | Part 1: Standard of Care
Number analyzed (Participants) | 19 | 19 | 22
PaO2/FiO2 ratio | 32.2 [-24.0 to 56.2] | 58.5 [10.1 to 150.4] | 7.5 [-14.7 to 33.5]
Statistical Analysis 1: Comparison: Part 1: Alteplase Low Dose vs Part 1: Standard of Care; Based upon Hedges-Lehmann estimator handling deaths as failure and Wilcoxon rank sum test methodology; Test type: Other; Median Difference (Net) = 17.193, 95% CI 2-sided [-28.45 to 52.33] — Calculated as alteplase dose group - standard of care alone
Statistical Analysis 2: Comparison: Part 1: Alteplase High Dose vs Part 1: Standard of Care; Based upon Hedges-Lehmann estimator handling deaths as failure and Wilcoxon rank sum test methodology; Test type: Other; Median Difference (Final Values) = 54.436, 95% CI 2-sided [0.49 to 110.36] — Calculated as alteplase dose group - standard of care alone

8. Secondary Outcome: Number of Oxygen-free Days up to Day 28
Description: Number of oxygen-free days (OFD) up to Day 28. Oxygen-free is defined as free from assistance from oxygen support. The number of oxygen-free days starts from when the patient has a 'lasting' value on the WHO clinical progression scale of ≤ 4 and ends on Day 28. A lasting value of ≤ 4 means that the value cannot exceed 4 at a later timepoint. If the patient is liberated from oxygen on Day x, then the number of OFDs is 28-x. If a patient has withdrawn consent prior to day 28 then he will have a missing value for OFD. In any case, if the status of the patient at Day 28 is death, as determined from the vital status page then the OFD=0.
Time Frame: Up to 28 days.
Population: Full Analysis Set (FAS) consisted of all randomised patients with at least one baseline and one post baseline assessment relating to the primary endpoint. The endpoint was only planned for subjects in Part 2.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Part 2: Alteplase High Dose - Non-invasive Mechanical Ventilation (NIV) Patients | Part 2: Standard of Care - Non-invasive Mechanical Ventilation (NIV) Patients | Part 2: Alteplase High Dose - Invasive Mechanical Ventilation (IMV) Patients | Part 2: Standard of Care - Invasive Mechanical Ventilation (IMV) Patients
Number analyzed (Participants) | 17 | 8 | 12 | 5
Days | 7.0 [0.0 to 20.0] | 4.5 [0.0 to 12.5] | 0.0 [0.0 to 5.5] | 0.0 [0.0 to 13.0]

9. Secondary Outcome: Length of Hospital Stay up to Day 28
Description: Length of hospital stay up to day 28 was determined based upon the first hospital discharge date, or discharge to another care facility. If the patient died within the first 28 day period, then length of hospital stay was 28.
Time Frame: Up to 28 days.
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Part 2: Alteplase High Dose - Non-invasive Mechanical Ventilation (NIV) Patients | Part 2: Standard of Care - Non-invasive Mechanical Ventilation (NIV) Patients | Part 2: Alteplase High Dose - Invasive Mechanical Ventilation (IMV) Patients | Part 2: Standard of Care - Invasive Mechanical Ventilation (IMV) Patients
Number analyzed (Participants) | 17 | 8 | 12 | 5
Days | 28.0 [16.0 to 28.0] | 24.0 [17.0 to 28.0] | 28.0 [26.0 to 28.0] | 28.0 [16.0 to 28.0]
Statistical Analysis 1: Comparison: Part 2: Alteplase High Dose - Non-invasive Mechanical Ventilation (NIV) Patients vs Part 2: Standard of Care - Non-invasive Mechanical Ventilation (NIV) Patients; Unadjusted mean difference: A restricted maximum likelihood (REML) based Analysis of Covariance (ANCOVA) was used. Adjustment was made for treatment; Test type: Other; p = 0.9856, ANCOVA; Median Difference (Net) = 0.1, 95% CI 2-sided [-7.5 to 7.6], Standard Error of Mean 3.6 — Calculated as alteplase dose group - standard of care alone
Statistical Analysis 2: Comparison: Part 2: Alteplase High Dose - Non-invasive Mechanical Ventilation (NIV) Patients vs Part 2: Standard of Care - Non-invasive Mechanical Ventilation (NIV) Patients; Adjusted mean difference: A restricted maximum likelihood (REML) based Analysis of Covariance (ANCOVA) was used. Adjustment was made for treatment, the number of days under NIV support, baseline D-Dimer level and age; Test type: Other; p = 0.8729, ANCOVA; Mean Difference (Net) = -0.6, 95% CI 2-sided [-8.5 to 7.3], Standard Error of Mean 3.8 — Calculated as alteplase dose group - standard of care alone

10. Secondary Outcome: Worst PaO2/FiO2 Ratio Change From Baseline to Day 6
Description: Worst PaO2/FiO2 ratio (or inferred PaO2/FiO2 ratio from SpO2) change from baseline to day 6. This assessment was planned to be measured on each of days 0 to 6. but only whilst the patients was still in hospital. The worst (lowest) daily measurement will be used and the higher the value the better the health status of the patient.
  * If the patient was still in hospital during day 6 then the day 6 value was used
  * If the patient was discharged from hospital prior to day 6 then the value at the time of hospital discharge was used
  * If the patient died prior to day 6 then the last value prior to death was used
  * If day 6 value was missing but Day 5 value available, the day 5 value was used
  * If day 6 value was missing, no Day 5 value available, but day 7 available, then day 7 value was used
  * Otherwise value was set to missing for that patient. Based upon this, the change from baseline for each patient was calculated and used for the analysis.
Time Frame: Up to 7 days.
Population: as for outcome 8
Measure: Mean (Standard Error); unit: PaO2/FiO2 ratio
Arm/Group | Part 2: Alteplase High Dose - Non-invasive Mechanical Ventilation (NIV) Patients | Part 2: Standard of Care - Non-invasive Mechanical Ventilation (NIV) Patients | Part 2: Alteplase High Dose - Invasive Mechanical Ventilation (IMV) Patients | Part 2: Standard of Care - Invasive Mechanical Ventilation (IMV) Patients
Number analyzed (Participants) | 17 | 8 | 12 | 5
PaO2/FiO2 ratio | 70.8 (20.7) | 0.0 (29.2) | -10.9 (13.1) | 3.4 (20.2)
Statistical Analysis 1: Comparison: Part 2: Alteplase High Dose - Non-invasive Mechanical Ventilation (NIV) Patients vs Part 2: Standard of Care - Non-invasive Mechanical Ventilation (NIV) Patients; [analysis description as in outcome 9, analysis 1]; Test type: Other; p = 0.0603, ANCOVA; Mean Difference (Net) = 70.9, 95% CI 2-sided [-3.3 to 145.1], Standard Error of Mean 35.8 — Calculated as alteplase dose group - standard of care alone
Statistical Analysis 2: Comparison: Part 2: Alteplase High Dose - Non-invasive Mechanical Ventilation (NIV) Patients vs Part 2: Standard of Care - Non-invasive Mechanical Ventilation (NIV) Patients; Adjusted mean difference: A restricted maximum likelihood (REML) based Analysis of Covariance (ANCOVA) was used. Adjustment was made for treatment, the number of days under NIV support, baseline D-Dimer level, baseline PaO2/FiO2 ratio and age; Test type: Other; p = 0.0362, ANCOVA; Mean Difference (Final Values) = 87.2, 95% CI 2-sided [6.3 to 168.0], Standard Error of Mean 38.5 — Calculated as alteplase dose group - standard of care alone

ADVERSE EVENTS:
Time Frame: From start of treatment (Alteplase) or randomisation (SOC) until the earliest of: Start point + 288 hours or last administration of Alteplase + 168 hours, up to 13 days.
Description: Treated Set (TS), included all patients who were randomised and, for patients in the alteplase groups, treated with at least one dose of trial drug.
Arm/Group | Part 1: Alteplase Low Dose | Part 1: Alteplase High Dose | Part 1: Standard of Care | Part 2: Alteplase High Dose - Non-invasive Mechanical Ventilation (NIV) Patients | Part 2: Standard of Care - Non-invasive Mechanical Ventilation (NIV) Patients | Part 2: Alteplase High Dose - Invasive Mechanical Ventilation (IMV) Patients | Part 2: Standard of Care - Invasive Mechanical Ventilation (IMV) Patients
All-Cause Mortality (participants affected / at risk) | 6/20 | 6/20 | 9/22 | 2/17 | 3/8 | 3/12 | 2/5
Serious Adverse Events (participants affected / at risk) | 8/20 | 10/20 | 12/22 | 7/17 | 4/8 | 9/12 | 2/5
Other Adverse Events (participants affected / at risk) | 11/20 | 11/20 | 12/22 | 12/17 | 4/8 | 11/12 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Alteplase Low Dose (N=20) | Part 1: Alteplase High Dose (N=20) | Part 1: Standard of Care (N=22) | Part 2: Alteplase High Dose - Non-invasive Mechanical Ventilation (NIV) Patients (N=17) | Part 2: Standard of Care - Non-invasive Mechanical Ventilation (NIV) Patients (N=8) | Part 2: Alteplase High Dose - Invasive Mechanical Ventilation (IMV) Patients (N=12) | Part 2: Standard of Care - Invasive Mechanical Ventilation (IMV) Patients (N=5)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Splenic infarction (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute right ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial injury (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0 | 1 | 0
Catheter site haemorrhage (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 1
Puncture site haemorrhage (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vessel puncture site haematoma (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic infarction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Device related bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 2 | 0 | 2 | 0 | 1 | 0
Pneumonia aspiration (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia pneumococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia staphylococcal (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 1 | 0 | 4 | 0 | 1 | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Traumatic lung injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vasoplegia syndrome (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 3 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1 | 1 | 1 | 2 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 6 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Alteplase Low Dose (N=20) | Part 1: Alteplase High Dose (N=20) | Part 1: Standard of Care (N=22) | Part 2: Alteplase High Dose - Non-invasive Mechanical Ventilation (NIV) Patients (N=17) | Part 2: Standard of Care - Non-invasive Mechanical Ventilation (NIV) Patients (N=8) | Part 2: Alteplase High Dose - Invasive Mechanical Ventilation (IMV) Patients (N=12) | Part 2: Standard of Care - Invasive Mechanical Ventilation (IMV) Patients (N=5)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 2 | 0 | 1 | 1
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Right ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 3 | 1 | 3 | 0 | 3 | 2
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Administration site haematoma (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Catheter site haemorrhage (General disorders) | 1 | 1 | 0 | 1 | 0 | 2 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Disease progression (General disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0
Hyperthermia (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1
Mucosal haemorrhage (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 2 | 0 | 0 | 1 | 1
Biliary dilatation (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aspergillus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Enterobacter infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Klebsiella bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neisseria infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 2 | 4 | 3 | 0 | 2 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 1 | 1 | 1 | 0 | 1
Pneumonia serratia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia staphylococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Stenotrophomonas infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Tracheobronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0 | 0 | 2 | 0 | 0
Vulvitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fibrin D dimer increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Glomerular filtration rate increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cell death (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 3 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0 | 2 | 1 | 1 | 2 | 0
Hyperlactacidaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2 | 3 | 1 | 0 | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aggression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 2 | 0 | 2 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0
Haemorrhage urinary tract (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oliguria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 0 | 2 | 0 | 2 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 2 | 0 | 2 | 0 | 0 | 0 | 2
Hypotension (Vascular disorders) | 0 | 1 | 1 | 2 | 1 | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Results for the invasive mechanical ventilation (IMV) patients were only analyzed descriptively due to insufficient enrolled patients. For the All-Cause Mortality endpoint, the non-invasive mechanical ventilation (NIV) arm did not have enough events to perform the adjusted statistical model, instead the unadjusted model is presented for this endpoint.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-02-17): https://cdn.clinicaltrials.gov/large-docs/94/NCT04640194/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-26): https://cdn.clinicaltrials.gov/large-docs/94/NCT04640194/SAP_001.pdf